CLINICAL TRIAL: NCT06512480
Title: Implementation in Colorectal Surgery of a New Modular and Open Robotic Platform.Pilot Project.
Brief Title: Colorectal Surgery, a New Robotic Platform (Hugo Ras)
Status: Recruiting | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Ana Sánchez Romero, GENERAL AND DIGESTIVE SURGEON, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: COLOROBOT-ELX24
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Surgery
Keywords: Robotic surgery; colorrectal surgery; Hugo™ RAS system; Surgical Innovations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PATIENTS UNDERGOING HUGO RAS COLORECTAL RESECTION: Patients will undergo colonic or colorectal resection with the Hugo RAS robotic platform.
  Interventions: Procedure: colonic resection

INTERVENTIONS:
Procedure: colonic resection — colonic resection with the Hugo RAS robotic platform.

SUMMARY:
A novel robotic platform -Hugo Robotic Assisted Surgery (RAS)- has been introduced with several innovations that may prove advantageous for surgeons such as an open console and four interchangeable modular arms. Our study aims to evaluate the safety, efficacy and potential impact of this platform in the surgical treatment of colorectal pathology.

DETAILED DESCRIPTION:
A case series underwent robotic-assisted colorectal procedures with the Hugo™ RAS system in General University Hospital of Elche, a referral center for colorectal surgery with extensive experience in laparoscopic surgery and none in robotics, from October 2023.No specific exclusion criteria were applied for patient selection. 2 surgeons and 1 nurse had previously completed the technical training [9] on the platform. The data were included in a computer database anonymously. For each patient, demographic, clinical and perioperative data, intraoperative robotics platform details, postoperative complications, length of hospital stay, tumor stage (TNM), and follow-up at one month were collected. For statistical analysisSPSS version 29.0 was used . In the descriptive analysis, the appropriate estimators have been used according to the type of variables: means or medians, standard deviation or ranges, for the quantitative variables, and percentages for qualitative variables.

Ethical approval was obtained from the ethical committee of the General University Hospital of Elche (PI 60/2024).

This study will be conducted in accordance with the Declaration of Helsinki on ethical principles for medical research on human subjects, which has its origin in the current review (revised version of Fortaleza, 2013) approved by the World Medical Assembly, the Oviedo Convention, and with the requirements current regulators included in the specific Spanish legislation: SAS order 3470/2009).

The rights, safety and well-being of study patients are the most important considerations to take into account and should prevail on the interests of science and society.

An informative document, Patient Information Sheet and Informed consent to patients to whom it is offered participate in the study. To be included in the study you must submit it signed and thus accepting the processing of your data and participation.

The processing, communication and transfer of personal data of all The participating subjects will comply with the current Organic Law 3/2018 of 5 December, Protection of personal data and guarantee of rights digital, adopting Regulation (EU) 2016/679 of the European Parliament and of the Council of April 27, 2016 on the protection of natural persons regarding the processing of your personal data and free circulation of these data and which repeals Directive 95/46/EC (General Regulation data protection), as well as Directive (EU) 2016/680 of the Parliament European Parliament and of the Council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data by of the competent authorities for the purposes of prevention, investigation, detection or prosecution of criminal offenses or execution of sanctions criminal offenses, and the free circulation of said data and repealing the Decision Framework 2008/977/JHA of the Council. The data collected for the study will be identified by a code, so in a manner that does not include information that could identify you, and only your doctor studio/collaborators may relate said data to you and your history clinic. Therefore, your identity will not be revealed to anyone except exceptions in case of medical emergency or legal requirement. The treatment, the communication and transfer of personal data of all Participants will comply with the provisions of this law. This study meets all the requirements regarding privacy of personal data. All Subsequent publication of results will never show data patient's personal. The data will be collected in an online database on the RedCap platform to establish a single and common registry of investigation responsibility of the institution and will be discussed within the framework of your participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Pacientes intervenidos de forma programada de procedimientos en cirugía colorrectal abdominal (neoplasia de colon, neoplasia de recto, diverticulosis, resección intestinal, cirugía transanal mínimamente invasiva (TAMIS), con la plataforma robótica Hugo™ RAS, en régimen de protocolos de rehabilitación multimodal (protocolos ERAS) (ANEXO 2).
* Edad mayor o igual a 18 años.

Exclusion Criteria:

* Pacientes intervenidos mediante abordaje inicial laparoscópico o abierto.
* Resecciones colorrectales de carácter urgente.
* Pacientes menores de 18 años.
* Existencia de otros procesos quirúrgicos concomitantes.
* Deterioro cognitivo severo que imposibilita la colaboración del paciente.
* Pacientes diagnosticados en estadio IV oncológico.
* Pacientes que rechacen participar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pacientes con indicación oncológica o de resección colónica.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-07-09 (Estimated); Study Completion 2027-07-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the results of a modular and open robotic platform (System of robotic-assisted surgery (RAS) Hugo™) in colorectal surgery (CRC) by complying with the quality indicators recommended by the Spanish Association of Coloproctology (AECP). | 1 year
  In the descriptive analysis, the appropriate estimators will be used according to the type of variables: means or medians, standard deviation (SD) or ranges, for the quantitative variables, and percentages (%) for qualitative variables. In the analysis bivariate, the Chi-square test will be used for qualitative variables, and for the quantitative variables the Student's t test if the distribution is normal and the Mann-Whitney U when such normality cannot be assumed (the normal distribution of the variables will be analyzed using the test of Kolmogorov-Smirnov).
  In all estimates, 95% confidence intervals will be calculated and a p value less than 0.05 will be considered significant.

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital of Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gueli Alletti S, Chiantera V, Arcuri G, Gioe A, Oliva R, Monterossi G, Fanfani F, Fagotti A, Scambia G. Introducing the New Surgical Robot HUGO RAS: System Description and Docking Settings for Gynecological Surgery. Front Oncol. 2022 Jun 9;12:898060. doi: 10.3389/fonc.2022.898060. eCollection 2022. PMID 35756633
- [Result] Bianchi PP, Salaj A, Rocco B, Formisano G. First worldwide report on Hugo RAS surgical platform in right and left colectomy. Updates Surg. 2023 Apr;75(3):775-780. doi: 10.1007/s13304-023-01489-5. Epub 2023 Mar 10. PMID 36897505
- [Result] Romero-Marcos JM, Sampson-Davila JG, Cuenca-Gomez C, Altet-Torne J, Gonzalez-Abos S, Ojeda-Jimenez I, Galaviz-Sosa ML, Delgado-Rivilla S. Colorectal procedures with the novel Hugo RAS system: training process and case series report from a non-robotic surgical team. Surg Endosc. 2024 Apr;38(4):2160-2168. doi: 10.1007/s00464-024-10760-8. Epub 2024 Mar 6. PMID 38448626
- [Result] Gangemi A, Bernante P, Rottoli M, Pasquali F, Poggioli G. Surgery of the alimentary tract for benign and malignant disease with the novel robotic platform HUGOTM RAS. A first world report of safety and feasibility. Int J Med Robot. 2023 Aug;19(4):e2544. doi: 10.1002/rcs.2544. Epub 2023 Jul 3. PMID 37395314
- [Result] Caruso R, Vicente E, Quijano Y, Ferri V. New era of robotic surgery: first case in Spain of right hemicolectomy on Hugo RAS surgical platform. BMJ Case Rep. 2023 Dec 28;16(12):e256035. doi: 10.1136/bcr-2023-256035. PMID 38154867
- [Result] Belyaev O, Fahlbusch T, Slobodkin I, Uhl W. Major colorectal surgery with Hugo RAS: initial experience of a German center and a review of the literature. Updates Surg. 2024 Sep;76(5):1705-1714. doi: 10.1007/s13304-024-01939-8. Epub 2024 Jul 9. PMID 38980596
- [Derived] Arroyo A, Lopez-de-Lerma C, Perea M, Sanchez-Romero A, Lopez-Rodriguez-Arias F, Alcaide MJ, Serrano-Navidad M, Barber X, Miranda E, Munoz-Rodes JL, Sanchez-Guillen L. Functional, oncologic and clinical outcomes of robotic rectal resection using the Hugo RAS system versus laparoscopic surgery: A comparative cohort study. Int J Colorectal Dis. 2026 Jan 22;41(1):40. doi: 10.1007/s00384-025-05063-w. PMID 41571968
- [Derived] Arroyo A, Sanchez-Romero A, Soler-Silva A, Quinto S, Lopez-Rodriguez-Arias F, Alcaide MJ, Serrano-Navidad M, Miranda E, Munoz JL, Sanchez-Guillen L. Utility guideline and considerations for the novel Hugo RAS (robotic-assisted surgery) system in colorectal surgery: surgical outcomes and initial experience in a tertiary center. Int J Colorectal Dis. 2024 Sep 18;39(1):144. doi: 10.1007/s00384-024-04715-7. PMID 39289218

DOCUMENTS (3):
  • Study Protocol (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT06512480/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT06512480/SAP_001.pdf
  • Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT06512480/ICF_002.pdf